CLINICAL TRIAL: NCT02050789
Title: Allowing Flexibility in Surgical Resident Duty Hours Trial
Brief Title: Flexibility In Duty Hour Requirements for Surgical Trainees Trial - "the FIRST Trial"
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American College of Surgeons (Other); American Board of Surgery (Other); Accreditation Council for Graduate Medical Education (Other)
Responsible Party: Principal Investigator, Karl Bilimoria, Assistant Professor of Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FIRST Trial
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Patient Safety; Resident Work Hours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Arm (No Intervention): Programs will continue adhering to current ACGME requirements.
- Intervention Arm (Experimental): The intent of the intervention arm is to allow flexibility in surgical resident duty hours and improve continuity of care.
  Interventions: Behavioral: flexible duty hours

INTERVENTIONS:
Behavioral: flexible duty hours — If a hospital is assigned to the intervention arm, all categorical and preliminary general surgery residents in that general surgery program will switch to the flexible duty hours while at an enrolled hospital.
  Other Names: Waiver from current duty hour requirements by the ACGME.; Allowed to eliminate all resident duty hour rules except:; Duty hours limited to 80 hrs/week averaged over 4 weeks.; Min of 1 free day (no duty)/week averaged over 4 weeks.; No in-house call > every 3rd night, averaged over 4 weeks.; Can increase chief residents duty requirements.
  Arms: Intervention Arm

SUMMARY:
Resident duty hour requirements in the U.S. are still evolving as stakeholders continue to debate how best to (re)structure postgraduate medical education.

There is concern that current restrictions may be detrimental to patient care and resident training. To investigate these issues, the investigators will be conducting a one-year, prospective randomized trial to examine how flexibility of duty hour requirements affects patient care when compared to current resident duty hour requirements. Further information about the study is available on the FIRST Trial website http://www.thefirsttrial.org/.

DETAILED DESCRIPTION:
Residency programs will be randomized to either (1) an intervention arm that eliminates several Accreditation Council for Graduate Medical Education (ACGME) duty hour requirements or (2) to a usual care arm where programs will continue adhering to current ACGME requirements. Programs in the intervention arm will be granted a waiver from current duty hour requirements by the ACGME and allowed to eliminate all resident duty hour rules with the following exceptions: Duty hours limited to 80 hours/week averaged over 4 weeks, minimum of one free day (no duty)/week averaged over 4 weeks, may not take in-house call more frequently than every 3rd night, averaged over 4 weeks, allowed to increase duty requirement flexibility for chief residents. The intent of the intervention arm is to allow flexibility in surgical resident duty hours and improve continuity of care. Subsequently, the investigators will compare multiple postoperative outcomes between the two study arms using data collected through the American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP). The results of this study will provide high-quality empirical evidence upon which to base resident duty hour requirements in the future.

Updated April 1, 2014

Detailed statistical analysis plan available on the FIRST Trial website. http://www.thefirsttrial.org/Approval/Approval

A listing of the 152 ACS-NSQIP hospitals that have elected to participate in the FIRST Trial is available on the FIRST Trial website. http://www.thefirsttrial.org/Hospitals/Hospitals

Updated July 14, 2014

Post-Randomization documents available for control and intervention arms on FIRST Trial website.

http://www.thefirsttrial.org/PostRandomization/PostRandomization

Updated August 2014

'FIRST Trial-Policies & Procedures Survey for Program Directors' survey administered to general surgery program directors via Survey Monkey.

Updated January 2015

Resident survey regarding duty hour policies and procedures administered at the end of the annual ABS In-Training Examination (ABSITE®).

Updated April 1, 2015

The Data Safety Monitoring Board (DSMB) was convened March 10, 2015 to review the results of planned interim analysis. After review, they voted to allow the FIRST Trial to continue. All other aspects of the trial are on track.

Updated May 24, 2016

Results from the study were released February 2, 2016 and the study has been extended for an additional year, through the 2016-2017 academic year.

Additional programs were enrolled in the one-year extension study.

March 10, 2017

The Accreditation Council for Graduate Medical Education (ACGME) released a final set of revisions to the professional standards all accredited US residency and fellowship programs follow in preparing today's physicians for a lifetime of practice. The new model also directly addresses requests from medical educators and residents by recognizing the risk of burnout and depression for physicians. Programs and institutions will be responsible for prioritizing physician well-being, ensuring protected time with patients, minimizing non-physician obligations, and ensuring that residents have the opportunity to access medical and dental care.

The total number of clinical and educational hours for residents has not changed. Starting the 2017-2018 academic year, the standards require that all programs and residents adhere to the maximum limits averaged over four weeks:

* a maximum of 80 hours per week
* one day free from clinical experience or education in seven
* in-house call no more frequent than every third night
* a maximum of 24 continuous work hours for all residents.

Updated September 12, 2017

Resident survey data collected with the 2016 and 2017 ABSITE Survey were collected and analyzed. Topics that emerged for further qualitative and quantitative analysis are as follows:

* Gender differences in resident outcomes
* Burnout and psychological wellbeing among residents
* Coercion and the decision to stay longer shifts within the flexible arm
* Needle stick and motor vehicle accident rates among US General Surgery residents
* Residency preparation (readiness) and the effects on burnout and wellbeing

ELIGIBILITY:
Inclusion Criteria:

* General Surgery Residency Programs participating in ACS NSQIP

Exclusion Criteria:

* Childrens' and VA Hospitals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Death or Serious Morbidity | 30 days
  The primary outcome for the trial is a composite measure of Death or Serious Morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Y. Bilimoria, MD MS, Principal Investigator — Northwestern University, American College of Surgeons

REFERENCES:
- [Derived] Saadat LV, Dahlke AR, Rajaram R, Kreutzer L, Love R, Odell DD, Bilimoria KY, Yang AD. Program Director Perceptions of Surgical Resident Training and Patient Care under Flexible Duty Hour Requirements. J Am Coll Surg. 2016 Jun;222(6):1098-105. doi: 10.1016/j.jamcollsurg.2016.03.026. Epub 2016 Apr 4. PMID 27234632
- [Derived] Bilimoria KY, Chung JW, Hedges LV, Dahlke AR, Love R, Cohen ME, Hoyt DB, Yang AD, Tarpley JL, Mellinger JD, Mahvi DM, Kelz RR, Ko CY, Odell DD, Stulberg JJ, Lewis FR. National Cluster-Randomized Trial of Duty-Hour Flexibility in Surgical Training. N Engl J Med. 2016 Feb 25;374(8):713-27. doi: 10.1056/NEJMoa1515724. Epub 2016 Feb 2. PMID 26836220
- [Derived] Bilimoria KY, Chung JW, Hedges LV, Dahlke AR, Love R, Cohen ME, Tarpley J, Mellinger J, Mahvi DM, Kelz RR, Ko CY, Hoyt DB, Lewis FH. Development of the Flexibility in Duty Hour Requirements for Surgical Trainees (FIRST) Trial Protocol: A National Cluster-Randomized Trial of Resident Duty Hour Policies. JAMA Surg. 2016 Mar;151(3):273-81. doi: 10.1001/jamasurg.2015.4990. PMID 26720622
- See also: Flexibility In duty hour Requirements for Surgical Trainees Trial - "The FIRST Trial" — http://www.thefirsttrial.org/